CLINICAL TRIAL: NCT05522621
Title: The Efficacy and Safety of Chinese Herbal Compound TJAOA102 in the Treatment of Menopausal Syndrome: A Multicenter, Prospective and Before-after Study.
Brief Title: A Muticenter Clinical Study of Chinese Herbal Compound TJAOA102 in Alleviating Menopausal Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shixuan Wang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220634-MS
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Menopausal Syndrome
Keywords: Menopausal Syndrome; Traditional Chinese Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJAOA102 (Experimental): Once enrolled, participants will be administrated TJAOA102 and followed by a 3-month medication cycle. The usage of this herbal compound is to take orally twice a day(two sacks per). Add it to about 200ml warm water and take it half an hour before breakfast in the morning and half an hour before bedtime in the evening except menstrual period.
  Interventions: Drug: TJAOA102

INTERVENTIONS:
Drug: TJAOA102 — Once enrolled, participants will be administrated TJAOA102

SUMMARY:
Currently, TCM recipes are widely used in treating menopausal syndrome(MS) with obvious efficiency and slight side effects. We have developed the Chinese herbal compound TJAOA102 and has validated its effects in animals. Here, we will perform a population-based, multicenter study to confirm the safety and efficacy of TJAOA102 in therapy of MS, which will provide a solid evidence for TCM in therapy of MS.

DETAILED DESCRIPTION:
Early menopause which is caused by DOR and POI may accelerate the aging of women, and lead to osteoporosis, cardiovascular and cerebrovascular diseases, frequent urination, dysuria, and decreased sleep quality. Postmenopausal women may suffer from osteoporosis and atherosclerosis, coronary heart disease and high blood pressure due to elevated cholesterol, triglycerides and low-density lipoproteins. Hence, the intervention for MS is indispensable. Currently, hormonotherapy(HT) is the first-line drug therapy recommended by clinical treatment guidelines. It can add exogenous sex hormones by replenishing the lack of hormones to relieve the symptoms caused by ovarian function decline, and then improve the health and life quality.However, HT also increased the risk of breast cancer, phlebothrombosis and so on. Hence, besides HT, TCM is an effective and alternative option.

To address this question, firstly we screened the database from the perspective of western medicine to identify the candidate Chinese herbs. Then multiple model organisms were used to verify their safety and effectiveness. Next, from the view of TCM, the pharmacological action, dose, synergistic effect and incompatibility were determined and finally TJAOA102, a Chinese medicine recipe for anti-ovarian aging was created. The essence of menopause is ovarian aging, so we developed anti-ovarian aging formula-TJAOA102.

At present, there is no guideline for long-term TCM management in treating MS. A clinical trial is imperative to test the safety and efficacy of TCM prescription. This study is a multicenter and prospective trial aiming to determine the safety and efficacy of TJAOA102 for preventing among women who were diagnosed with MS.

ELIGIBILITY:
Inclusion Criteria:

1. The age range of patient is 18-55 years old.
2. The diagnosis of women is DOR, POI, early menopause or menopausal syndrome, and wish to improve ovarian function or menopausal syndrome.
3. Sign the informed consent form.

Exclusion Criteria:

(1) The patient is known to be allergic or unsuitable for the Chinese herbal compound. (2) Women who are pregnant and lactating.

(3) Patients of POI or DOR had been menopause for more than 1 year. (4) Abnormal uterine bleeding, except ovulation disorders. (5) Women who is taking hormone drugs and has stopped taking them within 3 months; (6) The diagnosis of women is endometriosis, myadenosis, submucosal fibroids or the size of non-submucosal fibroids is more than 4 cm.

(7) The nature of pelvic mass is unknown. (8) The diagnosis of women is polycystic ovary syndrome, hyperprolactinemia, hyperandrogenemia, diabetes, thyroid and adrenal dysfunction and other endocrine diseases affecting ovulation.

(9) Patients with serious primary diseases such as cardiovascular, liver, kidney, lung, biliary, hematopoietic system (Hb<90g/L) and malignant tumor, and psychiatric patients.

(10) Patients who are participating in other clinical trials or have participated in other clinical trials within the last month.

(11) Patients who are unsuitable for the study evaluated by the investigator.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the change of Kupperman Index Score（KMI） | 6 months
  Assessing the KMI before and after the treatment of TJAOA102

SECONDARY OUTCOMES:
recovery rate of ovarian function | 6 months
  the recovery of ovarian function is defined as serum AMH increased more than 50%, or serum bFSH decreased more than 50%, or antral follicle count(AFC) increased more than 50% compared with that before treatment，or recover to normal level.